CLINICAL TRIAL: NCT03421678
Title: Ethnic/Racial Differences in Metabolism and DNA Adduct Formation by 1,3-butadiene
Brief Title: Ethnic/Racial Differences in Metabolism and DNA Adduct Formation
Status: Withdrawn | Type: Observational
Why Stopped: Study was completed at other sites
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017NTLS019
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Japanese American: Two parents of Japanese descent
  Interventions: Diagnostic Test: Urine Sample
- Non-Hispanic Whites: Two parents of non-Hispanic white descent
  Interventions: Diagnostic Test: Urine Sample
- Native Hawaiians: At least one parent of Hawaiian descent
  Interventions: Diagnostic Test: Urine Sample

INTERVENTIONS:
Diagnostic Test: Urine Sample — One to two home visits where tobacco use and medical history and biological samples will be collected including blood, buccal cells and urine

SUMMARY:
The study will investigate the role of 1,3-butadiene metabolic activation and deactivation in lung cancer risk among various ethnic/racial groups. This project will require urine samples from smokers and nonsmokers from the three ethnic/racial groups recruited by the Clinical and Biomarker Core for the analysis of 1,3-butadiene DNA adducts. Data on nicotine intake (urinary TNE) in these subjects as well as in 400 lung cancer cases and 400 controls from Project 1 will be also required for this project.

ELIGIBILITY:
Inclusion Criteria:

* One of the three targeted ethnic groups:

  * Japanese American - two parents of Japanese descent
  * Non-Hispanic Whites - two parents of non-Hispanic white descent
  * Native Hawaiians will include individuals with at least one parent of Hawaiian descent;
* Smoke 5 cigarettes per day over the past three months;
* >21 years of age;
* Consumes 14 or fewer drinks of alcohol per week;
* Generally stable and good health (determined by review of medical history);
* Able to provide written voluntary consent before performance of any study related procedure.

Exclusion Criteria:

* Current use of other nicotine containing products for > 4 times per month (and no use of any nicotine-containing products except cigarettes for 2 weeks prior to their study visits);
* Acute or uncontrolled medical or psychiatric conditions;
* Currently taking any medications that affect relevant metabolic enzymes or anti- inflammatory medications such as ibuprofen (this will be reviewed by study investigators on a case-by-case basis);
* Active infection (e.g., influenza, cold, respiratory infection, sinus infection) at the time of the visit;
* Pregnant or nursing or planning on becoming pregnant during the study;
* Unable to read and understand English.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 300 smokers will be recruited from the Multiethnic Cohort (MEC) study or the general population in Hawai'i
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Butadiene-DNA adducts in different ethnic groups | Day 1 & 2
  Investigate ethnic differences in butadiene-DNA adducts in smokers belonging to different ethnic groups.
Butadiene-DNA adduct load in smokers with lung cancer | Day 1 & 2
  Investigate the association between butadiene-DNA adduct load and lung cancer development in smokers.
Polymorphisms of carnicogen metabolizing genes | Day 1 & 2
  Examine how polymorphisms of carcinogen metabolizing genes influence metabolic inactivation, DNA adduct formation/repair, and toxicity of butadiene-derived epoxides.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — University of Minnesota, Department of Psychiatry